CLINICAL TRIAL: NCT00421486
Title: Incidence, Prevalence, Spectrum of HPV-types, and Viral Load Determination of High-risk Human Papillomavirus Infection of the Oral Cavity in HIV-infected Men Who Have Sex With Men
Brief Title: Oral Human Papillomavirus Infection in HIV-infected Men
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Deutsche Luft und Raumfahrt (Other Government)
Responsible Party: Principal Investigator, Alexander Kreuter, Prof. Dr., Deutsche Luft und Raumfahrt
Other Study IDs: 01 KI 0501
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Papillomavirus Infections; HIV Infections
Keywords: Oral human papillomavirus infection; HIV-infection; High-risk HPV viral load; Oral human papillomavirus infection in HIV-positive men; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — Papillomavirus Infections; HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Oral swabs for HPV-typing and high-risk HPV-determination — Oral swabs for HPV-typing and high-risk HPV-determination

SUMMARY:
Human papillomavirus (HPV)-infection belong to the most common sexually transmitted diseases worldwide. HIV-infected men having sex with men /MSM) are strongly associated with a higher prevalence of genitoanal HPV-infection, and perianal HPV-infections have been detected in up to 90% of HIV-positive men. The data concerning the incidence of oral HPV-infection in HIV-positive men, especially in the era of highly antiretroviral therapy, are conflicting. Thus, this prospective study mainly focuses on the incidence and prevalence of oral HPV-infection, spectrum of HPV-types, and oral high-risk HPV viral load in HIV-positive men.

DETAILED DESCRIPTION:
Human papillomavirus (HPV)-infection belong to the most common sexually transmitted diseases worldwide. Estimated prevalences of subclinical genital HPV-infection in the immunocompetent sexually active population range from 10 to above 50%. Genetic or iatrogenic immunosuppression is known to play a decisive role in the initiation of a variety of cutaneous neoplasias and their precursor lesions. In this context, HPV-associated anogenital malignancies occur with high frequency in patients with HIV-infection. In several studies, perianal HPV-infections have been detected in up to 90% of HIV-positive men and a high incidence of anal dysplasia has been reported in these patients. The data concerning the incidence of oral HPV-infection in HIV-positive men, especially in the era of highly antiretroviral therapy, are conflicting. Thus, this prospective study mainly focuses on the incidence and prevalence of oral HPV-infection, spectrum of HPV-types, and oral high-risk HPV viral load in HIV-positive men.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected men who have sex with men

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected men who have sex with men
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-03; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Spectrum of HPV types and associated clinical lesions | swabs will be obtained approximately every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kreuter, MD, Principal Investigator — Department of Dermatology, Ruhr University Bochum; Norbert Brockmeyer, MD, Principal Investigator — Department of Dermatology, Ruhr University Bochum; Ulrike Wieland, MD, Principal Investigator — Institute of Virology, University of Cologne
Locations (2):
- Germany (2):
  - Department of Dermatology, Ruhr University Bochum, Bochum, North Rhine-Westphalia
  - Institute of Virology, University of Cologne, Cologne, North Rhine-Westphalia

REFERENCES:
- See also: Deutsches Kompetenznetz HIV/AIDS — http://www.kompetenznetz-hiv.de